CLINICAL TRIAL: NCT01614808
Title: Observational - Characterization of Urinary Metabolite Profiles in Wilms Tumor
Brief Title: Studying Biomarkers in Urine Samples From Younger Patients With Wilms Tumor
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AREN12B7; NCI-2012-01973 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Recurrent Wilms Tumor and Other Childhood Kidney Tumors; Stage III Wilms Tumor
MeSH Terms: conditions — Wilms Tumor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: Archived urine samples are analyzed for specific metabolite patterns by nuclear magnetic resonance (NMR) spectroscopy and principal component analysis (PCA). Tumor tissue may also be examined by NMR and PCA.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research study is looking at biomarkers in urine samples from patients with Wilms tumor. Studying samples of urine from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer. It may also help doctors predict how patients will respond to treatment

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize the urinary metabolite signature of 10 stage III, favorable-histology, Wilms tumor patients from the Cooperative Human Tissue Network (CHTN) Databank, as distinct from 10 normal controls.

II. To characterize and compare the urinary metabolite profile in 50 randomly selected, stage III, favorable-histology, Wilms tumor patients enriched with an additional 30 stage III Wilms tumor patients who have relapsed.

III. To establish if the potential poor outcome (defined as relapse) in the favorable-histology group has a specific metabolite signature.

IV. To characterize the urinary metabolite signature of Wilms tumor in patients with unfavorable histology (diffuse anaplasia) and compare it to those with favorable histology.

OUTLINE:

Archived urine samples are analyzed for specific metabolite patterns by nuclear magnetic resonance (NMR) spectroscopy and principal component analysis (PCA). Tumor tissue may also be examined by NMR and PCA.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stage III, favorable-histology Wilms tumors and patients diagnosed with stage III, favorable-histology Wilms tumors who have relapsed

  * Tumor samples available from both groups
* Urine samples from the CHTN bank
* Control urine samples
* Urine samples from patients with unfavorable histology
* Not specified
* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with stage III, favorable-histology Wilms tumors and patients diagnosed with stage III, favorable-histology Wilms tumors who have relapsed.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2012-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Identification of metabolomic markers in urine that would assist in identifying higher risk of relapse of Wilms tumor in otherwise lower-risk stratified patients as assessed by NMR spectroscopy and PCA | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Maclellan, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States